CLINICAL TRIAL: NCT02668952
Title: The Impact of Low Chloride Containing Fluids on Acute Kidney Injury After Cardiopulmonary Bypass as Assayed by Urinary [TIMP2*IGFBP7]
Brief Title: Fluid Chloride and AKI in Cardiopulmonary Bypass
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Neal Gerstein, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-572
Record Dates: First submitted 2016-01-20; First posted 2016-01-29 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Saline Solution; Sodium Chloride; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline group (Active Comparator): 0.9% Normal Saline (0.9% Sodium Chloride) injection intravenously as needed. The amount administered (dosage, frequency, and duration) will be left to the clinical judgment of the attending physicians, and will follow usual patterns of use in cardiac surgery patients.
  Interventions: Drug: 0.9% Normal Saline (0.9% Sodium Chloride) injection
- Isolyte group (Experimental): Isolyte S (B Braun, Irvine CA) injection intravenously as needed. The amount administered (dosage, frequency, and duration) will be left to the clinical judgment of the attending physicians, and will follow usual patterns of use in cardiac surgery patients. Isolyte S is a prepackaged solution containing sodium chloride 0.53%, sodium gluconate 0.5%, sodium acetate trihydrate 0.37%, potassium chloride 0.037%, and magnesium chloride hexahydrate 0.03% w/v.
  Interventions: Drug: Isolyte S injection

INTERVENTIONS:
Drug: 0.9% Normal Saline (0.9% Sodium Chloride) injection
  Arms: Normal Saline group
Drug: Isolyte S injection
  Arms: Isolyte group

SUMMARY:
Acute kidney injury (AKI) is a potential complication of cardiac surgery. In animal models, excess exogenous Cl- ion in the bloodstream is associated with AKI. Normal saline IV fluid has higher levels of Cl- ion than the blood usually carries. An alternative IV fluid sold under the name Isolyte has lower Cl- ion levels. There is no literature comparing AKI outcomes in cardiac patients between patients receiving normal saline vs. Isolyte. The investigators propose to recruit and randomize 30 trial-completing cardiac surgery patients (up to 40 enrolled) into 2 study arms and compare renal outcomes.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a potential complication for patients undergoing cardiac surgery. AKI in post-cardiac surgery patients is associated with adverse outcomes, such as prolonged intensive care and hospital stay, diminished quality of life, increased long-term mortality, and an increased risk of chronic kidney disease requiring dialysis. The mortality in cardiac surgery patients with AKI severe enough to require renal replacement therapy (RRT) can be as high as 60%. One of the putative agents associated with AKI in animal models receiving crystalloid fluids for resuscitative interventions is excess exogenous chloride ion (Cl-). As compared to non-Cl- containing solutions in animal models, excess Cl- appears to lead to a hyperchloremic metabolic acidosis, increased renal vascular resistance, reduced renal blood flow, and reduced glomerular filtration rate - all of which are injurious to kidney function.

Historically, one of the most common balanced salt-solutions used in adult cardiac surgery has been 0.9% normal saline (NS), a crystalloid solution with 154 mmol/L of Cl-. This is much higher than physiologic plasma levels of 103 mmol/L. Isolyte, a less commonly used crystalloid solution, is much closer to physiologic levels at 98 mmol/L Cl-. In the context of cardiac surgery, there is no literature expressly comparing the effects of balanced crystalloid solution such as Isolyte versus NS on AKI incidence. There is a single trial examining a low-Cl- containing colloid solution in cardiac surgery that found less metabolic acidosis; however, AKI or markers of AKI were not measured outcomes in that lone trial, so it is not known whether low Cl- solution will have any effect on AKI risk in humans.

AKI results from a series of extremely complex cellular and molecular pathways involving endothelial, epithelial, inflammatory, and interstitial cells. The gold standard for identification and classification of AKI is dependent on serial serum creatinine (Scr) measurements, but this measurement can be unreliable during acute changes in kidney function. Recent studies have shown that tissue inhibitor of metalloproteinase (TIMP-2) performs better than existing markers for predicting the development of moderate or severe AKI (Kidney Disease: Improving Global Outcomes [KDIGO] stage 2 or 3) within 12 hours of sample collection. To further enhance the sensitivity of utilizing TIMP-2, the investigators plan on also measuring urinary insulin-like growth factor-binding protein 7 (IGFBP7). Along with TIMP-2, IGFBP7 is also an inducer of G1 cell cycle arrest, a key mechanism implicated in AKI.

This study will utilize the urinary [TIMP-2]*[IGFBP7] multiplicative product as a composite biomarker index to investigate the impact of intraoperative infusion of NS versus Isolyte on post-cardiac surgery renal function. This biomarker should identify patients at risk of imminent (within 12 hours) AKI KDIGO criteria.

Patients presenting for cardiac surgery are already quite ill often with multiple comorbidities. Acute kidney injury in this population is associated with significant morbidity and mortality. The available literature indicates that a fairly simple intervention could plausibly reduce the incidence of AKI, but it has not yet been examined in humans. Generating an evidence basis for it will substantially improve the safety of patients who need cardiac surgery. This intervention to reduce AKI may also then be applied to the broader non-cardiac surgery population as well.

ELIGIBILITY:
Inclusion Criteria:

* Planned on- or off-pump cardiac surgery including: bypass grafting, valvular procedures, congenital defect correction, and thoracic aortic procedures or a combination of these procedures

Exclusion Criteria:

* Emergency surgery
* Pregnancy
* Previous renal transplantation
* Documented moderate to severe acute kidney injury prior to enrollment (e.g. RIFLE-I or RIFLE-F/KDIGO stage 2 or 3)
* Patients already receiving dialysis (acute or chronic) or in imminent need of dialysis at time of enrollment
* Chronic kidney disease without baseline serum creatinine value obtained within 6 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02-04 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Gerstein, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Hospital, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of study results, qualified researchers may contact the PI for the deidentified dataset.

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline Group: 0.9% Normal Saline (0.9% Sodium Chloride) injection intravenously as needed. The amount administered (dosage, frequency, and duration) will be left to the clinical judgment of the attending physicians, and will follow usual patterns of use in cardiac surgery patients.
  0.9% Normal Saline (0.9% Sodium Chloride) injection
- Isolyte Group: Isolyte S (B Braun, Irvine CA) injection intravenously as needed. The amount administered (dosage, frequency, and duration) will be left to the clinical judgment of the attending physicians, and will follow usual patterns of use in cardiac surgery patients. Isolyte S is a prepackaged solution containing sodium chloride 0.53%, sodium gluconate 0.5%, sodium acetate trihydrate 0.37%, potassium chloride 0.037%, and magnesium chloride hexahydrate 0.03% w/v.
  Isolyte S injection
Period: Overall Study
Arm/Group | Normal Saline Group | Isolyte Group
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Saline Group | Isolyte Group | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (11.0) | 62.8 (9.4) | 64.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 10 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 30
[TIMP2] x [IGFBP7] [Mean (Standard Deviation); unit: (ng/mL)^2/1000] — This measure is an index consisting of the product of laboratory-derived serum concentrations of tissue inhibitor of metalloproteinase 2 and insulin-like growth factor binding protein 7.
  (ng/mL)^2/1000 | 0.101 (0.096) | 0.116 (0.138) | 0.108 (0.115)
Serum creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.93 (0.18) | 0.88 (0.14) | 0.91 (0.16)
Serum chloride [Mean (Standard Deviation); unit: mmol/L] | 108 (3.1) | 106 (3.4) | 107 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in [TIMP2]*[IGFBP7] Biomarker
Description: The difference in the [TIMP2]*[IGFBP7] biomarker between the preoperative value and a repeated measurement at 24 hours postoperatively. Positive values represent increase; negative values represent decrease
Time Frame: Baseline and postoperatively at 24 hours
Measure: Mean (Standard Deviation); unit: (ng/mL)^2/1000
Arm/Group | Normal Saline Group | Isolyte Group
Number analyzed (Participants) | 16 | 14
(ng/mL)^2/1000 | 0.015 (0.125) | 0.009 (0.148)

2. Secondary Outcome: Serum Creatinine Level at 24 Hours
Description: Serum creatinine measurement at 24 hours
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Normal Saline Group | Isolyte Group
Number analyzed (Participants) | 16 | 14
mg/dL | 0.85 (0.24) | 0.80 (0.16)

3. Secondary Outcome: Serum Chloride Level at 24 Hours
Description: Serum chloride ion measurement at 24 hours postoperatively
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Normal Saline Group | Isolyte Group
Number analyzed (Participants) | 16 | 14
mmol/L | 110 (3.0) | 106 (3.1)

4. Secondary Outcome: Proportion of Patients With Need for Dialysis
Description: Clinically-determined need for dialysis prior to discharge from hospital
Time Frame: One week
Measure: Number; unit: percentage of patients
Arm/Group | Normal Saline Group | Isolyte Group
Number analyzed (Participants) | 16 | 14
percentage of patients | 0 | 0

5. Secondary Outcome: Postoperative Arterial pH
Description: Arterial pH, measured 24 hours after surgery
Time Frame: One day
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Normal Saline Group | Isolyte Group
Number analyzed (Participants) | 16 | 14
pH | 7.38 (0.03) | 7.41 (0.05)

6. Secondary Outcome: Serum Creatinine Level at 48 Hours
Description: Serum creatinine level 48 hours postoperatively
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Normal Saline Group | Isolyte Group
Number analyzed (Participants) | 16 | 14
mg/dL | 0.91 (0.31) | 0.74 (0.14)

7. Secondary Outcome: Serum Chloride at 48 Hours
Description: Serum chloride measurement at 48 hours postoperatively
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Normal Saline Group | Isolyte Group
Number analyzed (Participants) | 16 | 14
mmol/L | 107 (4.6) | 104 (3.0)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Normal Saline Group | Isolyte Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-07): https://cdn.clinicaltrials.gov/large-docs/52/NCT02668952/Prot_SAP_000.pdf